CLINICAL TRIAL: NCT00005701
Title: Acute Cardiac Ischemia in Women in the ACI/TIPI Trial
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4301; R01HL053900 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2000-04

CONDITIONS: Heart Diseases; Cardiovascular Diseases; Angina Pectoris; Myocardial Ischemia
MeSH Terms: conditions — Heart Diseases; Cardiovascular Diseases; Angina Pectoris; Myocardial Ischemia

SUMMARY:
To conduct a series of five inter-related studies on acute cardiac ischemia (ACI) in women.

DETAILED DESCRIPTION:
BACKGROUND:

Acute cardiac ischemia (ACI), including acute myocardial infarction (AMI) and unstable angina pectoris, is the leading cause of death in women in the US. Despite growing interest in ischemic (coronary) cardiac disease in women, little research has focused on women in the most common site of ACI initial evaluation and care: the emergency department (ED). Improving medical care quality and outcomes for ACI in women will require an understanding of gender's influence on initial ED presentation, diagnosis, triage, treatment, and outcomes.The detail of prospectively-collected data and number of patients available for this project with the resulting large statistical power (while savings the cost of the $1.8 million ACI-TIPI Trial data collection effort) and the experience of the CCHSR in over a decade of related studies of factors influencing the triage, treatment, and outcome of ED patients with ACI, provide this project with substantial promise of new and useful results.

DESIGN NARRATIVE:

The five studies included. STUDY I: Were women's emergency department (ED) presentations of ACI different from men's? STUDY II: Were there differences between women and men in the ED diagnosis and triage of patients with chest pain and other symptoms suggestive of ACI? STUDY III: Were there differences between women and men in the use of non-invasive and invasive treatments among patients presenting to the ED with ACI? STUDY IV: Were there significant differences between women and men in medical outcomes during the acute event and within 30 days following ED presentation with ACI? STUDY V: Had differences between women and men in their ED presentation, diagnosis, and/or triage for chest pain or other symptoms compatible with ACI changed over the past 10-15 years? In studying the impact of gender, these studies also included analyses for primary and interaction effects related to patient sociodemographic features, ED presenting clinical features, physician type and training, hospital type and ED setting, health insurance type, and include adjustments for patients' probabilities of having ACI as well as their likelihood of acute cardiac mortality.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1994-07; Study Completion 1997-06 (Actual)

REFERENCES:
- [Background] Coronado BE, Griffith JL, Beshansky JR, Selker HP. Hospital mortality in women and men with acute cardiac ischemia: a prospective multicenter study. J Am Coll Cardiol. 1997 Jun;29(7):1490-6. doi: 10.1016/s0735-1097(97)00077-6. PMID 9180109
- [Background] Zucker DR, Griffith JL, Beshansky JR, Selker HP. Presentations of acute myocardial infarction in men and women. J Gen Intern Med. 1997 Feb;12(2):79-87. doi: 10.1046/j.1525-1497.1997.00011.x. PMID 9051556
- [Background] Maynard C, Beshansky JR, Griffith JL, Selker HP. Influence of sex on the use of cardiac procedures in patients presenting to the emergency department. A prospective multicenter study. Circulation. 1996 Nov 1;94(9 Suppl):II93-8. PMID 8901726